CLINICAL TRIAL: NCT02054377
Title: Cystic Fibrosis- Children and Adults Tai Chi Study: Can Tai Chi Improve Quality of Life for People With Cystic Fibrosis and Their Carers? Second Phase Study
Brief Title: Cystic Fibrosis- Children and Adults Tai Chi Study
Acronym: CFCATS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London South Bank University (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6463
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; tai chi
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (face to face tai chi) (Experimental): 1. 8 x 1 hour taught individual classes of Tai Chi over 3 months provided by a Tai Chi instructor at the participant's home/convenient location. These focus on 8 core postures. This is in addition to participant's usual routine care. A DVD and booklet to aid home practise will be provided.
  2. Daily home Tai Chi practise for 6 months (home practice encouraged for 5 to 10mins 5 times a week).
  3. At the end of the 9 months, local Tai Chi classes can be recommended if requested.
  Interventions: Other: Tai chi
- Group 2 (online tai chi) (Active Comparator): 1. 3 months usual routine care.
  2. 8 x 1 hour taught individual classes of Tai Chi over 3 months provided over the internet by a Tai Chi instructor. A DVD and booklet to aid home practise will be provided.
  3. Daily Tai Chi home practise for 6 months (home practice encouraged for 5 to 10mins 5 times a week).
  4. At the end of the 9 months, local Tai Chi classes can be recommended if requested.
  Interventions: Other: Tai chi

INTERVENTIONS:
Other: Tai chi — Tai Chi, a Chinese form of mindful exercise, may help alleviate CF symptoms, encourage active self-management and provide a practical way to relieve and manage stress for patients and carers. It involves gentle physical exercises, combined with breathing techniques and mindful awareness.
  It will be taught by qualified instructors either face to face in the participant's home or over videoconferencing technology e.g. Skype.
  A DVD of the Tai Chi was developed in Phase 1 which was successful for teaching adults, and will be used here, along with a child-friendly DVD. This will be filmed with and aimed at children aged 6-18. Teaching support materials, incorporating child-specific guidance such as animal-based Tai Chi movements, will be prepared for use in conjunction with the DVD.

SUMMARY:
Cystic fibrosis (CF) is a progressive disease. Symptoms include coughing, poor lung ventilation, recurrent infections, poor weight gain, diarrhoea, malnutrition, stress, frustration, depression, irritability, worry, insomnia, behavioural issues and missed school/work.

Tai chi, a Chinese form of exercise, uses slow choreographed movements, breathing exercises and mindfulness. Research suggests tai chi can improve physical and emotional wellbeing for various chronic conditions.

This study compares methods of teaching tai chi to 70 people with CF, and evaluates the effect on symptoms and quality of life. Adults and children with CF will be recruited and randomly allocated to an intervention group or a control group. The former will receive 8 individual face to face sessions of tai chi over a 3 month period and a video and handouts to aid home practice. The latter will have routine care for the first 12 weeks, followed by 8 individual online sessions of tai chi over a 3 month period, and a video and handouts for home practice.

Both groups will be encouraged to practice tai chi at home in the months following the taught sessions.

Questionnaire data on how participants and their carers are coping with CF, any general improvements in wellbeing, and differences in other clinical outcomes (medication etc.)will be collected. Data will be collected at the beginning and end of the intervention, and at 6 and 9 months post intervention and differences between the 2 groups compared over time.

Feedback from on line focus groups will ask about their experiences, feasibility of learning and practicing of tai chi, engagement with the process, perceived health impact, and experiences of participation.

It is hoped that the study may show how Tai Chi can help people with CF to maintain their health through mindful exercise, and improve troublesome symptoms like sleep and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CF
* no previous experience in Tai Chi, but ability/potential to undertake these movements
* able to commit to a 9 month study
* living in or near London or Brighton (depending on teacher locations)
* able to understand, read and write English
* 6 years old and above
* to have internet access for web based learning

Exclusion Criteria:

* participant in the feasibility phase
* currently taking part in another interventional research study

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cystic Fibrosis Questionnaire (CFQ-R ) | Change from baseline at 3 months
  • Cystic Fibrosis Questionnaire-Revised (CFQ-R), a disease-specific instrument (Quittner et al 2005; Modi & Quittner 2003). The CFQ uses 5 point Likert scales in 9 quality of life domains (physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions), 3 symptoms (weight, respiratory, and digestion) and health perception. CFQ-R was seen as acceptable, appropriate and easily completed in the feasibility study. There are four different versions of the CFQ-R which will be used as appropriate: Adult/adolescent version completed by the patient for those 14 and over; 12-13 year old version completed by the patient; parent CFQ for children aged 6 to 13; for children 6 to 11 child CFQ in interviewer format (parent/carer)
Cystic Fibrosis Questionnaire (CFQ-R ) | Change from baseline at 6 months
  • Cystic Fibrosis Questionnaire-Revised (CFQ-R), a disease-specific instrument (Quittner et al 2005; Modi & Quittner 2003). The CFQ uses 5 point Likert scales in 9 quality of life domains (physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions), 3 symptoms (weight, respiratory, and digestion) and health perception. CFQ-R was seen as acceptable, appropriate and easily completed in the feasibility study. There are four different versions of the CFQ-R which will be used as appropriate: Adult/adolescent version completed by the patient for those 14 and over; 12-13 year old version completed by the patient; parent CFQ for children aged 6 to 13; for children 6 to 11 child CFQ in interviewer format (parent/carer)
Cystic Fibrosis Questionnaire (CFQ-R ) | Change from baseline at 9 months
  • Cystic Fibrosis Questionnaire-Revised (CFQ-R), a disease-specific instrument (Quittner et al 2005; Modi & Quittner 2003). The CFQ uses 5 point Likert scales in 9 quality of life domains (physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions), 3 symptoms (weight, respiratory, and digestion) and health perception. CFQ-R was seen as acceptable, appropriate and easily completed in the feasibility study. There are four different versions of the CFQ-R which will be used as appropriate: Adult/adolescent version completed by the patient for those 14 and over; 12-13 year old version completed by the patient; parent CFQ for children aged 6 to 13; for children 6 to 11 child CFQ in interviewer format (parent/carer)

SECONDARY OUTCOMES:
Five facets mindfulness scale | Change from baseline at 3 months
  The five facets scale is a 39 item questionnaire about awareness of thoughts, anxieties, self-management
Five facets mindfulness scale | Change from baseline at 6 months
  The five facets scale is a 39 item questionnaire about awareness of thoughts, anxieties, self-management
Five facets mindfulness scale | Change from baseline at 9 months
  The five facets scale is a 39 item questionnaire about awareness of thoughts, anxieties, self-management

OTHER OUTCOMES:
Child and Adolescent Mindfulness Measure (CAMM) | Change from baseline at 3 months
  CAMM is a 10 item questionnaire about awareness of thoughts, anxieties, self-management.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline at 3 months
  Pittsburgh Sleep Quality Index (PSQI) (Buysse et al., 1989), a 10 item questionnaire about sleep quality and duration. This will be completed by the parent/carer for children under 12.
Routine clinical data from hospital records | Change from baseline at 3 months
  Changes in general health and respiratory function will be measured using routine clinical data from hospital records, to include: Body Mass Index (BMI), medications, antibiotic use, Forced Expiratory Volume (FEV1), Forced Vital Capacity (FVC), and oxygen saturation (amount of oxygen in red blood cells)
Modified Borg dyspnoea scale | Before and after each tai chi session
  Modified Borg dyspnoea scale is a one item, 10 point scale that rates comfort of breathing (American Thoracic Society, 2002, Borg and Borg, 2002, Borg, 1970)
Changes that week | Before and after each tai chi session
  Details of any changes in medication, exacerbations, antibiotic use, clinical trial participation, or care provision (start of session only), asked verbally by the instructor
Child and Adolescent Mindfulness Measure (CAMM) | Change from baseline at 6 months
  CAMM is a 10 item questionnaire about awareness of thoughts, anxieties, self-management.
Child and Adolescent Mindfulness Measure (CAMM) | Change from baseline at 9 months
  CAMM is a 10 item questionnaire about awareness of thoughts, anxieties, self-management.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline at 6 months
  Pittsburgh Sleep Quality Index (PSQI) (Buysse et al., 1989), a 10 item questionnaire about sleep quality and duration. This will be completed by the parent/carer for children under 12.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline at 9 months
  Pittsburgh Sleep Quality Index (PSQI) (Buysse et al., 1989), a 10 item questionnaire about sleep quality and duration. This will be completed by the parent/carer for children under 12.
Routine clinical data from hospital records | Change from baseline at 6 months
  Changes in general health and respiratory function will be measured using routine clinical data from hospital records, to include: Body Mass Index (BMI), medications, antibiotic use, Forced Expiratory Volume (FEV1), Forced Vital Capacity (FVC), and oxygen saturation (amount of oxygen in red blood cells)
Routine clinical data from hospital records | Change from baseline at 9 months
  Changes in general health and respiratory function will be measured using routine clinical data from hospital records, to include: Body Mass Index (BMI), medications, antibiotic use, Forced Expiratory Volume (FEV1), Forced Vital Capacity (FVC), and oxygen saturation (amount of oxygen in red blood cells)
Modified Borg dyspnoea scale | Change from baseline to 4 months
  Modified Borg dyspnoea scale is a one item, 10 point scale that rates comfort of breathing (American Thoracic Society, 2002, Borg and Borg, 2002, Borg, 1970)
Modified Borg dyspnoea scale | Change from baseline to 5 months
  Modified Borg dyspnoea scale is a one item, 10 point scale that rates comfort of breathing (American Thoracic Society, 2002, Borg and Borg, 2002, Borg, 1970)
Modified Borg dyspnoea scale | Change from baseline to 7 months
  Modified Borg dyspnoea scale is a one item, 10 point scale that rates comfort of breathing (American Thoracic Society, 2002, Borg and Borg, 2002, Borg, 1970)
Modified Borg dyspnoea scale | Change from baseline to 9 months
  Modified Borg dyspnoea scale is a one item, 10 point scale that rates comfort of breathing (American Thoracic Society, 2002, Borg and Borg, 2002, Borg, 1970)
Changes that week | Changes from baseline to 4 months
  Details of any changes in medication, exacerbations, antibiotic use, clinical trial participation, or care provision (start of session only), asked verbally by the instructor
Changes that week | Changes from baseline to 5 months
  Details of any changes in medication, exacerbations, antibiotic use, clinical trial participation, or care provision (start of session only), asked verbally by the instructor
Changes that week | Changes from baseline to 7 months
  Details of any changes in medication, exacerbations, antibiotic use, clinical trial participation, or care provision (start of session only), asked verbally by the instructor
Changes that week | Changes from baseline to 9 months
  Details of any changes in medication, exacerbations, antibiotic use, clinical trial participation, or care provision (start of session only), asked verbally by the instructor

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Robinson, PhD, Principal Investigator — LSBU
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Background] Ronan P, Mian A, Carr SB, Madge SL, Lorenc A, Robinson N. Learning to breathe with Tai Chi online - qualitative data from a randomized controlled feasibility study of patients with cystic fibrosis. Eur J Integr Med. 2020 Dec;40:101229. doi: 10.1016/j.eujim.2020.101229. Epub 2020 Oct 22. PMID 33106755
- [Background] Lorenc AB, Wang Y, Madge SL, Hu X, Mian AM, Robinson N. Meditative movement for respiratory function: a systematic review. Respir Care. 2014 Mar;59(3):427-40. doi: 10.4187/respcare.02570. Epub 2013 Jul 23. PMID 23882106
- [Background] Lorenc A, Ronan P, Mian A, Madge S, Carr SB, Agent P, Robinson N. Cystic fibrosis-Children and adults Tai Chi study (CF CATS2): Can Tai Chi improve symptoms and quality of life for people with cystic fibrosis? Second phase study protocol. Chin J Integr Med. 2015 May 26. doi: 10.1007/s11655-015-2150-1. Online ahead of print. PMID 26015075
- [Background] RONAN, P., MIAN, A., LORENC, A., CARR, S., MADGE, S. & ROBINSON, N. 2015b. CF-CATS2: Using technology to integrate Tai Chi into medical treatments for people with cystic fibrosis - An RCT. European Journal of Integrative Medicine, 7, Supplement 1, 47.
- [Background] RONAN, P., MIAN, A., LORENC, A., CARR, S., MADGE, S. & ROBINSON, N. 2015a. CF-CATS2: Is it feasible to use web-based technology to teach Tai Chi in order to integrate it into routine medical treatment for people with cystic fibrosis? European Journal of Integrative Medicine, 7, 693-694.
- See also: Information about the funder — http://www.tracielawlortrust.com/about-us/
- See also: Trailer for the study on you tube — http://youtu.be/eU5twohaSbE
- See also: Information about the funder — https://www.cysticfibrosis.org.uk/